CLINICAL TRIAL: NCT01997866
Title: Effects of Treating Sleep Apnea in Patients With Congestive Heart Failure
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Re-evaluate inclusion/exclusion criteria
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201300300
Record Dates: First submitted 2013-11-01; First posted 2013-11-28 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Obstructive Sleep Apnea; Sleep Apnea; Congestive Heart Failure; Heart Failure
Keywords: Obstructive Sleep Apnea; Sleep Apnea; Congestive Heart Failure; Heart Failure
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with Congestive Heart Failure (Other): STOP-BANG Scoring Model
  Polysomnogram Sleep Study
  Interventions: Other: STOP-BANG Scoring Model; Other: Polysomnogram Sleep Study

INTERVENTIONS:
Other: STOP-BANG Scoring Model — Patients with Congestive Heart Failure on non-Intensive Care Unit Medical Services and/or visiting our outpatient Congestive Heart Failure Clinic will be administered the STOP-BANG Scoring Model to determine whether they are considered high-risk or low-risk for Sleep Apnea.
Other: Polysomnogram Sleep Study — Patients determined by the STOP-BANG Scoring Model to be high-risk for Sleep Apnea will be referred to the Sleep Center physicians for evaluation and treatment. If medically indicated, a Polysomnogram Sleep Study will be performed.

SUMMARY:
Patients with Congestive Heart Failure (CHF) on non-Intensive Care Unit medical services and/or visiting our outpatient Congestive Heart Failure Clinic will be screened using the STOP-BANG Scoring Model. (STOP-BANG stands for Snoring, Tiredness, Observed Apnea, Blood Pressure, Body Mass Index, Age, Neck Circumference, Gender.) Patients with high risk of Obstructive Sleep Apnea (OSA) will be referred for evaluation and treatment of Sleep Apnea. They will be followed to determine if treatment of Sleep Apnea improves their quality of life and decreases their utilization of the Hospital and Emergency Department (ED).

DETAILED DESCRIPTION:
Patients with Congestive Heart Failure on non-Intensive Care Unit Medical Services and/or visiting our outpatient Congestive Heart Failure clinic will be screened using the STOP-BANG Scoring Model. Patients with high risk of Obstructive Sleep Apnea will be referred to the Sleep Center physicians for evaluation and treatment. Patients will be followed for one year to determine if the treatment for Sleep Apnea improves their Quality of Life and decreases Hospital and Emergency Department utilization.

ELIGIBILITY:
Inclusion criteria:

* Patient has:

  1. CHF (systolic, diastolic, any etiology), or
  2. Normal Ejection Fraction (EF) and most recent:

     1. Age less than 50: N-Terminal Pro Brain Natriuretic Peptide (NTPBNP) > 400,
     2. Age 50 and older: NTPBNP > 750,
     3. If no NTPBNP done: then Brain Natriuretic Peptide (BNP) > 200 (some newly referred patients will only have this available at their first visit, or
  3. Normal EF, no BNP done, and CHF documented in History or Problem List
* Admitted to the Hospital Medicine service, General Medicine Teaching service, Medicine Cardiology Team (MCT) service, Heart Failure service, or Community Health and Family Medicine (CHFM) service, OR Patient of the Congestive Heart Failure Clinic
* Patient has had at least 2 encounters (hospital inpatient admission, hospital observation admission, or ED visit) with University of Florida (UF) Health during the 12-month period immediately prior to the current admission (not including the current admission).
* English Speaking
* Males & Females
* Age 18 to 110
* Agreement to return to Gainesville for regular follow-up visits

Exclusion criteria:

* Decisionally impaired, cognitively impaired, or demented patient who has a surrogate, proxy, or guardian
* Current Drug/Alcohol abuse as evidenced by a) positive urine toxicology screen for cocaine or amphetamines during current admission, b) positive blood alcohol level upon admission, or c) documentation by current providers of continued abuse of alcohol or drugs
* Previous diagnosis of sleep apnea and on current treatment
* Uncontrolled Ventricular Dysrhythmias; sustained episodes of ventricular tachycardia or ventricular fibrillation in the hospital
* Evidence of current ischemia evidenced by elevated Troponin unrelated to Chronic Kidney Disease, or < 6 weeks since Myocardial Infarction (MI)
* Palliative care or Life expectancy < 6 months
* Isolated Cor Pulmonale - predominantly right ventricular dysfunction, Right Ventricular Systolic Pressure (RVSP) >50 and/or on the following medications for pulmonary hypertension: sildenafil (Viagra®), tadalafil (Adcirca®, Cialis®), IV or sub-cutaneous (SC) treprostinil (Remodulin®; Tyvaso™), ambrisentan (Letairis®), bosentan (Tracleer®), IV epoprostenol, inhaled iloprost (Ventavis®)
* On 5 liters or greater of O2
* Self-Pay Status
* Known Pregnancy
* Vulnerable Subjects such as prisoners, decisionally impaired/comatose individuals, terminally ill patients, UF/Shands/Veterans Administration (VA) staff, UF students

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Number of Hospital Admissions | Compare the number of Hospital Admissions during the 12-month period immediately prior to the index admission to the number of Hospital Admissions during the 12-month period immediately following the study intervention
Number of Hospitalized Days | Compare the number of Hospitalized Days during the 12-month period immediately prior to the index admission to the number of Hospitalized Days during the 12-month period immediately following the study intervention
Number of Emergency Department Visits | Compare the number of Emergency Department Visits during the 12-month period immediately prior to the index admission to the number of Emergency Department Visits during the 12-month period immediately following the study intervention

SECONDARY OUTCOMES:
Epworth Sleepiness Scale | Change from Baseline to 6 weeks
  Chance of Dozing Off - Scale: Never, Slight, Moderate, High
Epworth Sleepiness Scale | Change from Baseline to 12 months
  Chance of Dozing Off - Scale: Never, Slight, Moderate, High
Functional Outcome of Sleep Quality | Change from Baseline to 3 months
  Level of Difficulty Performing Everyday Activities - Scale: Don't do this activity, No difficulty, A little difficulty, Moderate difficulty, Extreme difficulty
Functional Outcome of Sleep Quality | Change from Baseline to 12 months
  Level of Difficulty Performing Everyday Activities - Scale: Don't do this activity, No difficulty, A little difficulty, Moderate difficulty, Extreme difficulty
Residual Apnea Hypopnea Index | at 6 weeks
  This is a data download from the Continuous Positive Airway Pressure machine, indicating the effectiveness of the patient's breathing while wearing the machine.
Epworth Sleepiness Scale | Change from Baseline to 3 months
  Chance of Dozing Off - Scale: Never, Slight, Moderate, High
Functional Outcome of Sleep Quality | Change from Baseline to 6 weeks
  Level of Difficulty Performing Everyday Activities - Scale: Don't do this activity, No difficulty, A little difficulty, Moderate difficulty, Extreme difficulty
Residual Apnea Hypopnea Index | at 3 months
  This is a data download from the Continuous Positive Airway Pressure machine, indicating the effectiveness of the patient's breathing while wearing the machine.
Residual Apnea Hypopnea Index | at 12 months
  This is a data download from the Continuous Positive Airway Pressure machine, indicating the effectiveness of the patient's breathing while wearing the machine.
% of nights with greater than 4 hours use of Continuous Positive Airway Pressure | at 6 weeks
  Compliance for a given night would be 4 hours use or more.
% of nights with greater than 4 hours use of Continuous Positive Airway Pressure | at 3 months
  Compliance for a given night would be 4 hours use or more.
% of nights with greater than 4 hours use of Continuous Positive Airway Pressure | at 12 months
  Compliance for a given night would be 4 hours use or more.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Leverence, M.D., Principal Investigator — University of Florida; Nila Radhakrishnan, M.D., Study Chair — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States